CLINICAL TRIAL: NCT03067233
Title: Automated Embedded Polysomnography
Brief Title: Automated Embedded Polysomnography (AEP)
Acronym: AEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ADOREPS_6
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2017-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polysomnography (Experimental): Three polysomnographic recordings will be made on 3 consecutive nights with Electroencephalogry.
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — Complete polysomnography with : Electroencephalogry, electro-oculography, surface electromyography (chin muscle, anterior tibial muscles), nasal pressure, respiratory movements (plethysmography of thoracic and abdominal inductance), pulse oximetry and electrocardiography.

SUMMARY:
To develop and validate a reliable automatic analysis of the signals recorded during a polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Insured by social security
* Speak french

Exclusion Criteria:

* Sleep disorder
* Neurologic, respiratory or cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the automatic analysis | 72 hour
  Comparison between polysomnographic analysis by two expert physicians and an automatic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Service des pathologies du sommeil - GH Pitié-Slapêtrière, Paris, France